CLINICAL TRIAL: NCT04240808
Title: Phase I Study of Feasibility and Safety of UCD19 Chimeric Antigen Receptor (CAR) T Cells in Adult Subjects With Relapsed/Refractory (R/R) B-Cell Non-Hodgkin's Lymphoma (B-NHL)
Brief Title: Study of Feasibility and Safety of UCD19 Chimeric Antigen Receptor (CAR) T Cells in Adult Subjects With Relapsed/Refractory (R/R) B-Cell Non-Hodgkin's Lymphoma (B-NHL)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 19-2807
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Non Hodgkin Lymphoma
Keywords: Car T; Car T Cells; Cancer; B-Cell Non-Hodgkin's Lymphoma; B-NHL
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms; Lymphoma, B-Cell

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- UCD19 CAR T Cells (Experimental): Participants will receive lymphodepleting chemotherapy followed by infusion of UCD19 CAR T Cells (Lentiviral Vector [LV] Transduced Autologous Peripheral Blood Lymphocytes
  Interventions: Biological: UCD19 CAR T Cells

INTERVENTIONS:
Biological: UCD19 CAR T Cells — Lymphodepleting chemotherapy followed by infusion of UCD19 CAR T Cells (Lentiviral Vector [LV] Transduced Autologous Peripheral Blood Lymphocytes)

SUMMARY:
This study will test whether immune cells modified to recognize B-cell non-Hodgkin lymphoma (NHL) can be successfully manufactured at the University of Colorado Anschutz and whether these cells can be administered with an acceptable safety profile. Adults who have been diagnosed with B-cell non-Hodgkin lymphoma (NHL) that has relapsed or no longer responds to chemotherapy (relapsed or refractory) may be eligible to participate in this study.

The investigators will use participants own immune cells, called T cells, to kill the lymphoma. These T cells are involved in fighting infections and in some cases, can also kill cancer cells. The investigators will extract T cells from the participant's blood, modify the cells in a laboratory, and then return teh cells to the participant's body via intravenous (IV) injection. In the laboratory, the investigators will add a new gene into the T cells that allows the T cells to recognize and kill the lymphoma cells, and allows these modified cells to multiply and increase in numbers. To put the new gene into your T cells, the investigators will use a weakened virus. The virus is modified so that it cannot multiply or spread once the cells are infused.

DETAILED DESCRIPTION:
The objective of this Phase 1 open-label study is to assess the feasibility of UCD19 Chimeric Antigen Receptor (CAR) T Cells manufacture onsite, successful infusion of eligible subjects, and safety of UCD19 CAR T Cells infusion in subjects with relapsed/refractory B-Cell Non-Hodgkin's Lymphoma (B-NHL).

Six (6) subjects will participate in the initial cohort of this open-label, single arm, single site study to assess dose-limiting toxicity (DLT) and safety; the first set of 3 subjects will initiate treatment with lymphodepleting chemotherapy prior to CAR T cell infusion staggered 30 days from CAR T cell dosing of the previously treated subject. Depending on the assessment of DLTs, the second set of 3 subjects may be enrolled and dosed without stagger.

After the initial 6 subjects have received treatment, an additional 14 subjects will participate in the Phase 1 expansion study.

Participants will include adults with relapsed/ primary refractory CD19 positive (i.e. CD19 expressing) B-NHL as confirmed by either flow cytometry, immunohistochemistry (IHC), or both who are not candidates for other curative forms of therapy. Enrolled participants will receive lymphodepleting chemotherapy followed by infusion of UCD19 CAR T Cells (Lentiviral Vector [LV] Transduced Autologous Peripheral Blood Lymphocytes). Participants will be enrolled up to 1 month before anticipated date of apheresis, and will be considered completed at 12 months post-treatment.

Long Term Follow Up will be conducted under a separate protocol and will occur for up to 15 Years to collect data on the long-term safety of UCD19 CAR T Cells, and for the observation, detection, and evaluation of latent adverse reactions including secondary malignancies.

While this study focuses on primary endpoints for feasibility of the manufacturing and infusion processes and safety of the administered UCD19 CAR T Cells, preliminary evidence of effectiveness will be collected and analyzed for use in planning future CAR T cell therapy studies.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated Informed Consent form.
* Stated willingness to comply with all study procedures and availability for the duration of the parent study and the long-term follow-up observational study.
* Male or non-pregnant, non-lactating females, aged 18 to 80 years.
* Performance status according to the Eastern Cooperative Oncology Group ≤ 2.
* Failed two or more lines of systemic therapy.
* Unable to receive commercially available CD19 CAR T Cells.
* Relapsed or primary refractory CD19 positive (i.e. CD19 expressing) B-NHL of the following types as confirmed by either flow cytometry, Immunohistochemistry (IHC), or both:

  * Diffuse large B-cell lymphoma (DLBCL)
  * Burkitt lymphoma
  * Intermediate lymphoma between Burkitt and DLBCL
  * Primary Mediastinal B-cell lymphoma (PMBL)
  * Follicular lymphoma
  * Mantle cell lymphoma (MCL)
  * Marginal zone lymphoma (MZL)
* No available curative alternative treatment, as determined by primary treating oncologist.
* No active Graft-versus-Host Disease (GvHD).
* In women of childbearing potential, willingness to use effective means of birth control for 1 year after UCD19 CAR T Cell infusion.

Exclusion Criteria:

* Prior therapies:

  * Received monoclonal antibody therapy within 14 days of the apheresis; or
  * Received immunomodulatory drugs (lenalidomide, tyrosine kinase inhibitors) within 14 days of the apheresis; or
  * Received corticosteroids more than 7.5mg/day within 14 days of the apheresis (physiologic replacement allowed up until apheresis, as clinically indicated); or
  * Allogeneic hematopoietic stem cell transplant with 90 days (immunosuppressive therapy for at least 4 weeks) of apheresis; or
  * Donor lymphocyte infusion within 4 weeks of apheresis.
  * Cluster of differentiation 3 (CD3) count <0.15 x 106 cells/mL
* Severe psychiatric illness that could impede the patient's ability to provide informed consent and/or adhere to the parent protocol and/or the long-term follow-up protocol.
* Active HIV (Acquired Immune Deficiency Syndrome) or history of HIV infection, as directed by schedule or if known.
* Active Hepatitis B or Hepatitis C infection.
* Diffusion capacity of the lungs for carbon monoxide < 40% predicted prior to lymphodepletion.
* Left ventricular ejection fraction < 40% (evaluated by echocardiogram [ECHO] or Multigated Acquisition Scan [MUGA]) prior to lymphodepletion.
* Transaminases > 5x upper limit of normal prior to lymphodepletion.
* Serum Bilirubin > 4 mg/dL prior to lymphodepletion.
* Serum Creatinine > 1.6 mg/dL or measured creatinine clearance < 50 mL/min prior to lymphodepletion.
* Active infection that is unresponsive to antimicrobial therapy prior to lymphodepletion.
* Females planning to become pregnant during the course of the study.
* Unwillingness or inability to comply with study visits and study procedures for the entire duration of study participation.
* Unsuitable for cellular therapy for any reason, in the opinion of the Investigator.
* Any prior gene therapy, including prior CAR T cell therapy.
* Active central nervous system (CNS) disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2020-07-17 (Actual); Primary Completion 2023-03-24 (Actual); Study Completion 2023-10-23 (Actual)

PRIMARY OUTCOMES:
Feasibility: Successful manufacture of UCD19 CAR T Cells, as determined by the number of successfully manufactured doses | Day 0 (infusion)
  The successful manufacture of UCD19 Chimeric Antigen Receptor (CAR) T Cells onsite meeting the IND-defined release criteria. Manufacture of UCD19 CAR T Cells will begin after enrollment and be completed within 1 month. Success will be determined by whether or not the participant's CAR T Cell count meets the target dose required for infusion at Day 0. The number of successfully manufactured doses will be reported.
Feasibility: Percent of Participants successfully infused with UCD19 CAR T Cells | Day 0 (infusion)
  The percent of participants who are able to receive an infusion of UCD19 CAR T cells.
Safety: Number of Participants Who Experience a Dose Limiting Toxicity (DLT) within 30 days after treatment | Up to 30 Days Post-Infusion
  The number of subjects who receive UCD19 CAR T Cells and experience a DLT within 30 days after treatment, as defined herein using the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5.0).
Safety: Percent of Participants Who Experience a Dose Limiting Toxicity (DLT) within 30 days after treatment | Up to 30 Days Post-Infusion
  The percent of all subjects who receive UCD19 CAR T Cells and experience a DLT within 30 days after treatment, as defined herein using the National Cancer Institute's (NCI) Common Terminology Criteria for Adverse Events (CTCAE v5.0).

SECONDARY OUTCOMES:
Efficacy: Overall response rate (Complete Response (CR)/Partial Response (PR)/Stable Disease (SD)) at 90 days | 90 Days Post-Infusion
  The number of participants with Complete Response (CR)/Partial Response (PR)/Stable Disease (SD) at 90 days post-treatment, as determined by the investigators.
Efficacy: Overall response rate (Complete Response (CR)/Partial Response (PR)/Stable Disease (SD)) at 6 Months | 6 Months Post-Infusion
  The number of participants with Complete Response (CR)/Partial Response (PR)/Stable Disease (SD) at 6 months post-treatment, as determined by the investigators.
Efficacy: Overall response rate (Complete Response (CR)/Partial Response (PR)/Stable Disease (SD)) at 1 Year | 1 Year Post-Infusion
  The number of participants with Complete Response (CR)/Partial Response (PR)/Stable Disease (SD) at 1 Year post-treatment, as determined by the investigators.
Efficacy: Rate of participants with Complete Response at 6 Months | 6 Months Post-Infusion
Efficacy: Rate of participants with Complete Response at 1 Year | 1 Year Post-Infusion
Efficacy: Median Duration of Remission at 1 Year | 1 Year Post-Infusion
Efficacy: Progression Free Survival (PFS) at 1 Year | 1 Year Post-Infusion
  Number of participants with Progression Free Survival (PFS) at 1 year post-infusion.
Efficacy: Overall Survival (OS) at 1 Year | 1 Year Post-Infusion
  Number of participants surviving at 1 year post-infusion.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Verneris, MD, Study Director — University of Colorado Denver, Anschutz Medical Campus; Manali Kamdar, MD, Principal Investigator — University of Colorado Denver, Anschutz Medical Campus
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No